CLINICAL TRIAL: NCT01132703
Title: A Phase I Randomized, Double-Blind, Placebo-Controlled Study to Assess the Safety, Tolerability, and Pharmacokinetics of Escalating Doses of RP-1127 (Glyburide for Injection) in Healthy Male and Female Volunteers
Brief Title: Safety Study of RP-1127 (Glyburide for Injection) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RPI 101
Record Dates: First submitted 2010-04-14; First posted 2010-05-28 (Estimated); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Traumatic Brain Injury; Stroke
MeSH Terms: conditions — Brain Injuries, Traumatic; Stroke | interventions — Glyburide; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Matching Placebo (Placebo Comparator): Matching placebo (glyburide excipients without active) is administered as a bolus followed by continuous infusion for 72 hours.
  Interventions: Drug: Placebo
- Glyburide for Injection: Dose 1 (Experimental): Glyburide is administered as a bolus followed by a infusion for 72 hours
  Interventions: Drug: Glyburide for Injection
- Glyburide for Injection: Dose 2 (Experimental): Glyburide is administered as a bolus followed by a infusion for 72 hours
  Interventions: Drug: Glyburide for Injection
- Glyburide for Injection: Dose 3 (Experimental): Glyburide is administered as a bolus followed by a infusion for 72 hours.
  Interventions: Drug: Glyburide for Injection

INTERVENTIONS:
Drug: Glyburide for Injection — Administered as specified in the Treatment Arm.
  Other Names: RP-1127; glibenclamide; glybenclamide
  Arms: Glyburide for Injection: Dose 1; Glyburide for Injection: Dose 2; Glyburide for Injection: Dose 3
Drug: Placebo — Administered as specified in the Treatment Arm.
  Arms: Matching Placebo

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of different dose levels of glyburide for injection, administered as a bolus dose followed by a 3-day continuous infusion. The secondary objectives are to assess the pharmacokinetics (PK) of glyburide and blood glucose and serum insulin pharmacodynamic (PD) responses to glyburide.

DETAILED DESCRIPTION:
This study was previously posted by Remedy Pharmaceuticals, Inc. and has since been acquired by Biogen.

ELIGIBILITY:
Inclusion Criteria:

1. A healthy male or a healthy nonpregnant, nonlactating female.
2. Capable of understanding and complying with the protocol and has signed the informed consent form before the Screening procedures begin.
3. Have a body mass index of between 18.0 and 30.0 kg/m², inclusive.
4. A clinically normal physical examination, 12-lead electrocardiogram (ECG), screening laboratory studies and urinalysis.
5. A negative urine or saliva test for selected substances of abuse and cotinine.

Exclusion Criteria:

1. Clinically significant history of hypoglycemia as assessed by the investigator.
2. History of seizure disorder, even if currently not receiving anticonvulsant medications.
3. History of adverse reaction to glyburide, other sulfonylurea class of anti-diabetic medications, or other sulfa drugs.
4. Glucose-6-phosphate dehydrogenase (G6PD) deficiency as determined by G6PD enzyme testing at screening.
5. Be an active smoker or user of other forms of tobacco. Former smokers or tobacco users must have refrained from smoking or using other forms of tobacco for at least 6 months prior to dosing on Study Day 1.
6. A history or clinical manifestations of significant metabolic (including diabetes mellitus, hypercholesterolemia, or dyslipidemia), hematologic, pulmonary, cardiovascular, gastrointestinal, neurologic, hepatic, renal, urologic, immunologic, or psychiatric disorders (a history of mild depression, currently not receiving therapy, is acceptable).
7. Use any prescription medication within 14 days prior to randomization, or nonprescription drugs within 7 days. Exceptions may be made by the medical monitor on a case-by-case basis.
8. Received another investigational drug within 30 days prior to randomization.
9. A positive hepatitis virus test (Hepatitis B virus surface antigen or hepatitis C virus antibody) or a positive human immunodeficiency virus (HIV) antibody test at screening. If the HIV test is positive, the subject will be informed privately and referred for additional counseling.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2010-01-07 (Actual); Primary Completion 2010-05-07 (Actual); Study Completion 2010-05-07 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events and Serious Adverse Events | Up to Day 28
  An adverse event (AE) is defined as any untoward medical occurence such as a sign, symptom, and/or laboratory finding that is concurrent with the use of a drug in humans. A serious adverse event is any AE that is fatal, life-threatening, requires or prolongs hospital stay, results in persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event

SECONDARY OUTCOMES:
Pharmacokinetic (PK) Parameter of Glyburide: Clearance (CL) | Day 1 (baseline) and at multiple time points up to Day 5
PK Parameter of Glyburide: Volume of Distribution (Vz) | Day 1 (baseline) and at multiple time points up to Day 5
PK Parameter of Glyburide: Elimination Rate Constant (λz) | Day 1 (baseline) and at multiple time points up to Day 5
PK Parameter of Glyburide: Half-Life (t1/2) | Day 1 (baseline) and at multiple time points up to Day 5
PK Parameter of Glyburide: Predicted Steady-State Concentration (Css) | Day 1 (baseline) and at multiple time points up to Day 5
PK Paramater of Metabolites (M1 and M2): Maximum Plasma Concentrations (Cmax) | Day 1 (baseline) and at multiple time points up to Day 5
Pharmacodynamic (PD) Parameter of Glyburide: Change from Baseline in Blood Glucose | Day 1 (baseline) and at multiple time points up to Day 5
PD Parameter of Glyburide: Change from Baseline in Serum Insulin | Day 1 (baseline) and at multiple time points up to Day 5

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Jasper Clinic, Kalamazoo, Michigan, United States